CLINICAL TRIAL: NCT02423252
Title: The Effects of a Psycho-cognitive Nursing Intervention on Clinical and Psychological Outcomes of Critically Ill Patients: A Randomized Controlled Trial
Brief Title: Effects of a Psycho-cognitive Nursing Intervention on Patients' Outcomes in Critical Illness
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr Elizabeth Papathanassoglou (Other)
Collaborators: Nicosia General Hospital (Other)
Responsible Party: Sponsor-Investigator, Dr Elizabeth Papathanassoglou, Professor, Cyprus University of Technology
Organization: Cyprus University of Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EX 043 - EP1; EX 043 EPPSY-13 (Other Grant/Funding Number: Grant:Cyprus University of Technology/Funding number: EX 043)
Record Dates: First submitted 2015-03-28; First posted 2015-04-22 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Critical Illness; Stress; Inflammatory Response
Keywords: Critical illness; Intervention; RCT; Relaxation; Guided imagery; Touch/Massage; Music listening; Neuropeptides; Inflammatory molecules; Post-traumatic stress; Critical care nurse; Psychocognitive nursing intervention; Interpersonal support
MeSH Terms: conditions — Critical Illness | interventions — Massage; Imagery, Psychotherapy; Standard of Care

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Intervention: Massage, Relaxation, imagery, music. Patients in Intervention group will receive standard care plus massage, relaxation, guided imagery and music listening
  Interventions: Behavioral: Massage, Relaxation, Guided imagery and music listening.; Other: No Intervention
- Control (No Intervention): Patients in control group will receive standard care only. Same records and outcome measures with intervention group will apply for control group as well.

INTERVENTIONS:
Behavioral: Massage, Relaxation, Guided imagery and music listening. — In addition to standard care, patients in the intervention group will receive a 60 minutes individually delivered programme, administered once per day by a nurse (the researcher) for up to 5 days during staying in ICU. This session aims to induce relaxation and involves interpersonal support, touch/massage and through a headphone system relaxation and guided imagery exercises and music listening. Patients are provided a CD of the relaxation instructions, after their discharge, for own use
  Other Names: body-mind intervention
  Arms: Intervention group
Other: No Intervention — The control group will receive the standard care which includes the routine standard care provided by nurses, physiotherapists and intensivists or specialists (e.g. surgeons)
  Other Names: standard care, control
  Arms: Intervention group

SUMMARY:
The purpose of this study is to investigate whether a psycho-cognitive nursing intervention including relaxation, guided imagery, touch and music listening can improve the clinical and psychological outcome of critically ill patients. The investigators hypothesize that, patients who receive the proposed psycho-cognitive nursing intervention will report lower stress, less pain and have altered level of stress neuropeptides in peripheral blood, lower levels of inflammatory molecules, less complications and better self reported lived experience than patients who receive standard care alone.

DETAILED DESCRIPTION:
In previous research on the impact of stress on physiology, it has been shown that stress and its molecules may contribute to derangements prevalent in critical illness, including systemic inflammation, cellular stress, oxidative damage, endothelial dysfunction and coagulopathies which precipitate high mortality and morbidity. Investigators will examine whether a Psycho-cognitive nursing intervention to induce relaxation can improve patients outcomes.

Sixty ICU patients with or without SIRS will be randomized to receive either standard care or a brief Psycho-cognitive Nursing Intervention, plus standard care, up to 5 days during ICU stay.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients
* Understand Greek language
* Age over 18 years
* They have Richmond Agitation Sedation Scale rate: -3 +3
* Have an Arterial line in place

Exclusion Criteria:

* Patient who is expected to stay less than 24 hours in Critical care unit
* Have history of psychiatric disturbances
* Their condition does not permit use of headphones
* Have hearing impairment
* Receive neuro-muscular blockers
* Are confused
* Patients under universal conduct precautions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-11 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Change in Pain intensity [10-point numeric rating scale (NRS) scale] | from baseline to 60 min over 1-5 days. (baseline: just before 1st day starting intervention time).
Change in Pain intensity [Behavioral pain scale (BPS) scale] | from baseline to 60 min over 1-5 days. (baseline: just before 1st day starting intervention time).
Change in Pain intensity [critical-care pain observation tool (CPOT) scale] | from baseline to 60 min over 1-5 days. (baseline: just before 1st day starting intervention time).
Change in Systolic blood pressure (SBP) | from baseline to 30 and 60 min (baseline: just before 1st day starting intervention time), over 1 to 5 days.
Change in self reported Relaxation/calm levels (self- reported, 10 points NRS scale) | from baseline to 60 min (baseline: just before 1st day starting intervention time), over 1 to 5 days.
Change in Plasma Neuropeptide Y level | from baseline to 60 min (baseline: morning before 1st day intervention) (1st sample), morning after 1st day intervention (2nd sample), morning before and after intervention (1st and 2nd sample) on days 3rd and 5th.] [Designated as safety issue: No]
Change in Plasma Neuropeptide oxytocin level | from baseline to 60 min (baseline: morning before 1st day intervention) (1st sample), morning after 1st day intervention (2nd sample), morning before and after intervention (1st and 2nd sample) on days 3rd and 5th.] [Designated as safety issue: No]
Change in Plasma Neuropeptide beta-endorphin level | from baseline to 60 min (baseline: morning before 1st day intervention) (1st sample), morning after 1st day intervention (2nd sample), morning before and after intervention (1st and 2nd sample) on days 3rd and 5th.] [Designated as safety issue: No]
Change in Plasma Neuropeptide acetylcholine level | from baseline to 60 min (baseline: morning before 1st day intervention) (1st sample), morning after 1st day intervention (2nd sample), morning before and after intervention (1st and 2nd sample) on days 3rd and 5th.] [Designated as safety issue: No]
  Investigators will study the differences of clinical and biochemical parameters between randomized groups of patients treated and not treated with the intervention.
  Differences in levels of neuropeptides and inflammatory markers among patient groups (intervention group and comparison) and group of healthy volunteers.

SECONDARY OUTCOMES:
Change in Diastolic blood pressure (DAP) | from baseline to 30 and 60 min (baseline: just before 1st day starting intervention time), over 1 to 5 days.
Change in Mean arterial pressure (MAP) | from baseline to 30 and 60 min (baseline: just before 1st day starting intervention time),
Change in Heart rate (HR) | from baseline to 30 and 60 min (baseline: just before 1st day starting intervention time),
  Differences in levels of neuropeptides and inflammatory markers among patient groups (intervention group and comparison) and group of healthy volunteers.
Change in Respiration rate (RR) | from baseline to 30 and 60 min (baseline: just before 1st day starting intervention time),
Change in Temperature (TMP) | from baseline to 30 and 60 min (baseline: just before 1st day starting intervention time),
Sequential organ failure assessment (SOFA) scores | once on days 1, 3, 5 and on last day of stay in ICU.
Multiple organ disfunction syndrome (MODS) scores | once on days 1, 3, 5 and on last day of stay in ICU.
Self reported quality of Sleep [10-point numeric rating scale (NRS) scale] | morning before starting intervention (days 1-5)
Change in Self reported anxiety level [10-point numeric rating scale (NRS) scale] | from baseline to 60 min over 1-5 days. (baseline: just before 1st day starting intervention time).
Change in Self reported fear level [10-point numeric rating scale (NRS) | from baseline to 60 min over 1-5 days. (baseline: just before 1st day starting intervention time).
Change in Self reported optimism level [10-point numeric rating scale (NRS) | from baseline to 60 min over 1-5 days. (baseline: just before 1st day starting intervention time).
Change in Self reported distress level [10-point numeric rating scale (NRS)] | from baseline to 60 min over 1-5 days. (baseline: just before 1st day starting intervention time).
Richmond agitation-sedation scale (RASS) score | days 1, 2, 3, 4, 5.
Change in Plasma levels of Inflammatory marker Interleukin-6 | from baseline to 60 min (baseline: morning before 1st day intervention) (1st sample), morning after 1st day intervention (2nd sample), morning before and after intervention (1st and 2nd sample) on days 3rd and 5th.] [Designated as safety issue: No]
Change in Plasma levels of Inflammatory marker Interleukin-8 | from baseline to 60 min (baseline: morning before 1st day intervention) (1st sample), morning after 1st day intervention (2nd sample), morning before and after intervention (1st and 2nd sample) on days 3rd and 5th.] [Designated as safety issue: No]
Change in Plasma levels of Inflammatory marker soluble fas ligand (sfas) | from baseline to 60 min (baseline: morning before 1st day intervention) (1st sample), morning after 1st day intervention (2nd sample), morning before and after intervention (1st and 2nd sample) on days 3rd and 5th.] [Designated as safety issue: No]
Change in Plasma inflammatory marker levels High mobility group box-1 (HMGB-1)] | from baseline to 60 min (baseline: morning before 1st day intervention) (1st sample), morning after 1st day intervention (2nd sample), morning before and after intervention (1st and 2nd sample) on days 3rd and 5th.] [Designated as safety issue: No]
  Investigators will study the differences of clinical and biochemical parameters between randomized groups of patients treated and not treated with the intervention.
  Differences in levels of neuropeptides and inflammatory markers among patient groups (intervention group and comparison) and group of healthy volunteers.
assessment of psychological distress (ICUESS: Intensive Care Unit Environmental Stressor Scale, self-assessment in a 1-10 numerical analogue scale). | within 48 hours post discharge from ICU
Assessment of symptoms of post traumatic stress disorder (PTSD) using DTS (Davidson Trauma Scale) | one month and six months after hospital discharge
assessment of quality of life using Short Form 36 version2 scale (SF36v2) | one month and six months after discharge
Exploration of lived experience of critical illness (phenomenological interviews) | one month and six months after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth DE Papathanassoglou, Phd, Study Director — Cyprus University of Technology
Locations (1):
- Nicosia General Hospital, Nicosia, Cyprus